CLINICAL TRIAL: NCT02576769
Title: Melanocyte Features and Its Influence in Pigmentation in Basal Cell Carcinoma in the Mexican Population
Brief Title: The Role of Melanocyte in Basal Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo-Cazares, Study Director, Universidad Autonoma de San Luis Potosí
Other Study IDs: BCC1
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal cell carcinoma; Pigmentation; Melanocyte; Melanin; Skin cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Basal cell carcinoma: Basal cell carcinoma
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Basal cell carcinoma (BCC) is the most frequent neoplasia worldwide. There are more than 30 histopathologic subtypes, however the nodular subtype is the most common. Pigmented varieties are common in darker skin types, therefore in our country. Previous studies have shown an increase number and size of melanocytes. Melanogenesis were increased at the expense of hyperfunctioning melanocytes as well. The aim of the study was to describe the characteristics of melanocytes in pigmented and non-pigmented variants of basal cell carcinoma.

DETAILED DESCRIPTION:
Melanocytes are highly specialized dendritic cells that performs multiple functions through autocrine, paracrine and endocrine mechanisms. These cells are part of a complex system of intercellular communication along with keratinocytes, Langerhans cells and fibroblasts. This intricate network of cellular communication is possible thanks to interaction with cytokines, growth factors and neurotransmitters. Although melanocytes perform brilliantly immunoregulatory and neuroendocrine functions, their fundamental role is to offer protection against the harmful effects of UV radiation through production and transference of melanin to keratinocytes, a process better known as melanogenesis. The latter requires 3 basic proteins to ensure photoprotection: MC1R (activation), MITF (traduction) and TYR (melanin synthesis).

If one of the main features of melanocytes is to avoid UV radiation injurious effect, thus it raises many questions regarding the possible relation between these cells and skin cancer. Currently a great number of melanocytic alterations have been described in melanoma; however in non-melanoma skin cancer the role of melanocytes is less clear. Basal cell carcinoma (BCC) is the most frequent neoplasia worldwide. There are more than 30 histopathologic subtypes, however the nodular subtype is the most common. Pigmented varieties are common in darker skin types, therefore in our country. Previous studies have shown an increase number and size of melanocytes. Melanogenesis were increased at the expense of hyperfunctioning melanocytes as well. In our experience we have noticed the clinical course regarding pigmented nodular basal cell carcinoma is more benign when compared to those without pigment. Most studies regarding the role of melanocytes and pigmentation in basal cell carcinoma have been conducted in caucasian populations, and therefore not representative of what may occur in mestizo population. The aim of the study was to describe the characteristics of melanocytes in pigmented and non-pigmented variants of basal cell carcinoma. Quantify the expression of melanocytic maturation: transcription factors (SOX9 and SOX10), focal adhesion kinase (FAK125) and receptor tyrosine kinase (c-KIT) and melanogenesis such as melanocortin 1 receptor (MC1R), microphthalmia-associated transcription factor (MITF) and tyrosinase (TYR) markers. Investigate the tumoral microenvironment through the quantification of melanin, mast cells, angiogenesis and solar elastosis.

ELIGIBILITY:
Inclusion Criteria:

* Mexican subjects
* Age between 40 and 90 years
* Both genders
* Sign informed consent

Exclusion Criteria:

* Sign informed consent withdrawal

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with histologic diagnosis of basal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Melanocyte number | Up to 1 year
  To quantify the number of melanocytes in basal cell carcinoma
Melanocyte phenotype | Up to 1 year
  To quantify melanocyte maturation stages in basal cell carcinoma through markers
Melanogenesis characteristics | Up to 1 year
  To quantify the expression of melanogenic markers in basal cell carcinoma

SECONDARY OUTCOMES:
Melanin presence | Up to 1 year
  To quantify melanin deposition in basal cell carcinoma using special histologic stains (Fontana-Masson)
Vessels number (angiogenesis) | Up to 1 year
  To quantify number of vessels in basal cell carcinoma using special histologic stains (Elastic fibers)
Mast cells number | Up to 1 year
  To quantify melanocytes in basal cell carcinoma using special histologic stains (Giemsa)
Solar elastosis quantity | Up to 1 year
  To quantify solar elastosis in basal cell carcinoma using special histologic stains (Elastic fibers)

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Castanedo-Cazares, MD, MSc, Study Director — Hospital Central "Dr. Ignacio Morones Prieto"; Bertha Torres-Alvarez, MD, Study Chair — Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Lao LM, Kumakiri M, Kiyohara T, Kuwahara H, Ueda K. Sub-populations of melanocytes in pigmented basal cell carcinoma: a quantitative, ultrastructural investigation. J Cutan Pathol. 2001 Jan;28(1):34-43. doi: 10.1034/j.1600-0560.2001.280104.x. PMID 11168750
- [Background] Sakuraba K, Hayashi N, Kawashima M, Imokawa G. Down-regulated PAR-2 is associated in part with interrupted melanosome transfer in pigmented basal cell epithelioma. Pigment Cell Res. 2004 Aug;17(4):371-8. doi: 10.1111/j.1600-0749.2004.00156.x. PMID 15250939
- [Background] Frey LM, Houben R, Brocker EB. Pigmentation, Melanocyte Colonization, and p53 Status in Basal Cell Carcinoma. J Skin Cancer. 2011;2011:349726. doi: 10.1155/2011/349726. Epub 2010 Sep 29. PMID 21152129